CLINICAL TRIAL: NCT02436265
Title: Low Dose IV Dexamethasone in Prolonging Caudal Anesthesia in Children Undergoing Genitourinary Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment/lack of potential subjects fitting criteria
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Aali M. Shah, Aali Shah, MD, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1408968524
Record Dates: First submitted 2015-02-05; First posted 2015-05-06 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Surgery
Keywords: Neuraxial; Caudal; Block; Anesthesia; Dexamethasone
MeSH Terms: conditions — Bites and Stings | interventions — Dexamethasone; Calcium Dobesilate; Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Ropivacaine (Sham Comparator): Group 1 Ropivacaine Intervention: Each patient will receive a caudal with 1ml/kg of 0.2% ropivacaine
  Interventions: Drug: Ropivacaine
- Group 2 Ropivacaine and Dexamethasone (Active Comparator): Group 2 Ropivacaine/dexamethasone Intervention: Each patient will receive a caudal with 1ml/kg of 0.2% ropivacaine and 0.1mg/kg of intravenous dexamethasone immediately after caudal placement
  Interventions: Drug: Dexamethasone; Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexamethasone — IV dexamethasone
  Other Names: IV Decadron
  Arms: Group 2 Ropivacaine and Dexamethasone
Drug: Ropivacaine — Ropivacaine only
  Other Names: Ropi

SUMMARY:
Caudal injection of local anesthetic is a neuraxial technique routinely performed on young children for postoperative analgesia after lower abdominal and lower extremity surgical procedures. One of the major limitations of the use of single shot neuraxial injections for this purpose is the limited duration of action of the injected local anesthetic. Adjuvant medications, such as clonidine and epinephrine, have been added to the local anesthetic to prolong the duration of the neuraxial block, with varying results. Dexamethasone is a synthetic glucocorticoid steroid commonly used in the perioperative setting for a multitude of indications, including the prolongation of local anesthetic based analgesia. It has been shown that the administration of dexamethasone either intravenously or via perineural injection can significantly increase the duration of analgesia derived from a local anesthesia based peripheral nerve block. Literature also suggests that the effect of dexamethasone is equivalent whether given intravenously or perineurally. Interest in dexamethasone enhanced caudal analgesia exists and a previous study noted that caudal anesthesia can be prolonged by intravenous dexamethasone. The study was criticized for using a higher dose of dexamethasone (0.5 mg/kg) than is routinely used in the pediatric population outside of airway procedures, which may expose patients to dose related side effects of dexamethasone. A large meta-analysis has suggested that 0.1 mg/kg is effective for analgesic prolongation, but no direct study of low dose intravenous dexamethasone in combination with caudal anesthesia has been performed.

DETAILED DESCRIPTION:
As dexamethasone is an inexpensive and commonly used medication, it would be beneficial to know if a similar prolongation of analgesia occurs when a local anesthetic is given neuraxially in combination with low dose intravenous dexamethasone. This project will investigate the efficacy of low dose intravenous (IV) dexamethasone in prolonging the duration of post operative analgesia provided by an intraoperative caudal injection of local anesthetic. All patients will be enrolled in the study the day of surgery, in the preoperative waiting area. The study will be explained by an anesthesiologist with extensive knowledge of the protocol. Computer randomization will occur for each patient. Randomization will not increase the risk to either group as all medications and techniques utilized for this study are commonly accepted for routine care for these patients.

ELIGIBILITY:
Inclusion Criteria:

* age 2 to 10 years
* Scheduled for elective inpatient genitourinary surgical procedure
* Caudal anesthesia standard of care for surgical procedure
* have provided parental consent and assent in accordance with the institutional review board requirements

Exclusion Criteria:

* Abnormal/difficult anatomy
* known allergy to ropivacaine or dexamethasone
* history of documented chronic pain
* existing infection at site of intended injection

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2015-02; Primary Completion 2017-06-23 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aali M Shah, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Desmet M, Braems H, Reynvoet M, Plasschaert S, Van Cauwelaert J, Pottel H, Carlier S, Missant C, Van de Velde M. I.V. and perineural dexamethasone are equivalent in increasing the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder surgery: a prospective, randomized, placebo-controlled study. Br J Anaesth. 2013 Sep;111(3):445-52. doi: 10.1093/bja/aet109. Epub 2013 Apr 15. PMID 23587875
- [Background] Hong JY, Han SW, Kim WO, Kim EJ, Kil HK. Effect of dexamethasone in combination with caudal analgesia on postoperative pain control in day-case paediatric orchiopexy. Br J Anaesth. 2010 Oct;105(4):506-10. doi: 10.1093/bja/aeq187. Epub 2010 Jul 20. PMID 20659915
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 Ropivacaine | Group 2 Ropivacaine and Dexamethasone
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ropivacaine Only Group: Patients receiving caudals with local anesthetic, but no IV dexamethasone
- Ropivaciane + IV Dexamethasone: Patients receiving caudals with local anesthetic +0/1mg/kg IV dexamethasone
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Only Group | Ropivaciane + IV Dexamethasone | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 3 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Scores Over 24 Hours
Description: Will track the trend of pain scores for both arms to note differences in pain score based on intervention received. Pain scores will be based on a patient verbal response of 0-10 pain, 0 being no pain and 10 being worst pain, or with a FLACC score (Face, Legs, Activity, Cry, Consolability scale) of 0-10 if patient unable to communicate verbally
Time Frame: 24 hours
Population: The study was abandoned/terminated. Enrollment in the trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results. No participants were analyzed.
Groups:
- Ropivacaine Only: caudal analgesia with 0.2% ropivacaine only
- Ropivaciane + IV Dexamethasone: Caudal analgesia with IV dexamethasone
Arm/Group | Ropivacaine Only | Ropivaciane + IV Dexamethasone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Ropivacaine + IV Dexamethasone: Caudal analgesia with 0.2% ropivacaine only plus IV dexamethasone 0.1 mg/kg
Arm/Group | Ropivacaine Only | Ropivacaine + IV Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

LIMITATIONS AND CAVEATS:
The study was abandoned/terminated. Enrollment in the trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results. No participants were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT02436265/Prot_SAP_000.pdf